CLINICAL TRIAL: NCT02961257
Title: Randomized Multicenter, Phase III Trial Evaluating the Safety of 2 Schedules of Cabazitaxel (Bi-weekly Versus Tri-weekly) Plus Prednisone in Elderly Men (≥ 65years) With mCRPC Previously Treated With a Docetaxel-containing Regimen
Brief Title: Trial Evaluating the Safety of 2 Schedules of Cabazitaxel in Elderly Men With mCRPC Previously Treated With a Docetaxel
Acronym: CABASTY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Association Pour La Recherche des Thérapeutiques Innovantes en Cancérologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABASTY
Record Dates: First submitted 2016-08-22; First posted 2016-11-10 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2019-05

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — cabazitaxel; XRP6258; Prednisone; Granulocyte Colony-Stimulating Factor; Lenograstim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Cabazitaxel 25 mg/m² intravenously over 1 hour on Day 1of a 3-week cycle, plus prednisone (or prednisolone) 10 mg orally given daily for a maximum of 10 cycles (ie 30 weeks of treatment).
  Prophylactic Granulocyte colony-stimulating factor G-CSF (Granocyte) will be injected from Day 3 to Day 7 after every administration of cabazitaxel.
  Interventions: Drug: cabazitaxel; Drug: Prednisone; Drug: Granulocyte colony-stimulating factor (G-CSF)
- Arm B (Experimental): Cabazitaxel 16 mg/m2 on Day 1 and Day 15 of a 4-week cycle plus prednisone (or prednisolone) 10 mg per day up to 10 cycles (ie 40 weeks of treatment). Prophylactic Granulocyte colony-stimulating factor G-CSF (Granocyte) will be injected from Day 3 to Day 7 after every administration of cabazitaxel.
  Interventions: Drug: cabazitaxel; Drug: Prednisone; Drug: Granulocyte colony-stimulating factor (G-CSF)

INTERVENTIONS:
Drug: cabazitaxel — * Arm A : cabazitaxel 25 mg/m² on Day 1 of a 3-week cycle plus daily prednisone or
  * Arm B: cabazitaxel 16 mg/m² on Day 1 and Day 15 of a 4-week cycle plus daily prednisone.
  * Treatment will be continued for a maximum of 10 cycles unless there is documented disease progression or unacceptable toxicity.
  * Standard cabazitaxel premedication will be used
  Other Names: Jevtana; XRP6258
Drug: Prednisone — Arm A:plus prednisone 10 mg orally given daily for a maximum of 10 cycles Arm B: plus prednisone 10 mg orally given per day up to 10 cycles
Drug: Granulocyte colony-stimulating factor (G-CSF) — Primary prophylaxis with Granulocyte Colony-Stimulating Factor (G-CSF) will be injected from Day 3 to Day 7 after every administration of cabazitaxel
  Other Names: Granocyte

SUMMARY:
The purpose of this study is to evaluate the incidence of grade ≥ 3 neutropenia and/or neutropenic complications (febrile neutropenia, neutropenic infection) with two schedules of cabazitaxel (bi-weekly versus tri-weekly) plus prednisone in elderly men (≥ 65 years) with mCRPC previously treated with a docetaxel-containing regimen.

DETAILED DESCRIPTION:
Randomized, open-label, phase 3 trial in mCRPC patients aged ≥ 65 years.

Number of subjects:

Total:170 to 200 (85 to 100 per arm)

Treatment:

* Arm A : cabazitaxel 25 mg/m² on Day 1 of a 3-week cycle plus daily prednisone or
* Arm B: cabazitaxel 16 mg/m² on Day 1 and Day 15 of a 4-week cycle plus daily prednisone.
* Treatment will be continued for a maximum of 10 cycles unless there is documented disease progression or unacceptable toxicity.
* Standard cabazitaxel premedication will be used
* Prophylactic G-CSF (GRANOCYTE) will be injected from Day 3 to Day 7 after every administration cycle of cabazitaxel· All new hormonal treatment, including ODM-201, prior to study entry is allowed.
* Patients who received Radium-223 are eligible for this study
* Treatment with LHRH should not be discontinued.

Exploratory assessments:

CT-Scan (abdominal/pelvic/chest) or whole body MRI and Bone scan: at screening, every 3 months and EOT.

FACT-P questionnaire:at C1D1,each subsequent visit and EOT

Exploratory substudy Blood samples will be collected in France (4 or 6 sites) and the Netherlands (2 sites). Biomarker analysis will be conducted at the Urology and The Tumor Immunology Laboratory at Radboud UMC in NL.

Biomarker schedule Arm A (25mg/m2): Baseline - Week 6 - Week 12 - at progression Arm B (16mg/m2): Baseline - Week 6 - Week 12 - at progression Optional sample points are at C1D8.

Number of subjects: 50

Statistical analysis:

A sample size of 77 to 90 evaluable patients per arm will achieve 80% power to detect a 20% difference in G3 neutropenia incidence between the 2 arms. The incidence in group cabazitaxel 25 mg/m2 q3w is assumed to be 32% and 12% on bi-weekly cabazitaxel arm. The test used is a two-sided Fisher's exact test at 0.05 significance level. Assuming 10% non-evaluable patients, 85 to 100 patients should be included in each arm for a total of 170 to 200.

Patients will be stratified according to G8 score (< 14 vs. ≥ 14), and age (< 70 vs. ≥ 70) before randomization.

Exploratory sub-study The trial is powered on a clinical endpoint, namely to detect a 20% difference in G3 nThe trial is powered on a clinical endpoint, namely to detect a 20% difference in G3 neutropenia incidence between arms (32% in arm A vs 12% arm B; power 80% with two-sided alpha of 5%, correcting for 10% non-evaluable patients (=17 patients).

From the 153 to 180 evaluable patients, we have 76 to 90 patients in each arm, of which we expect 40-60 evaluable patients for translational studies (calculations performed on 25 per arm).

In arm A, we expect 8 patients (32% of patients) with G3 neutropenia, and 17 patients that do not. In arm B, we expect 3 patients (12% of patients) with G3 neutropenia, and 22 patients that do not. For the MDSC analyses, we therefore will be comparing 11 patients with G3 neutropenia to 39 patients.

For all continuous variables, including all immune subpopulations present in blood, mean (sd) will be presented if the distribution seems to be symmetric and in case of a skewed distribution the median and IQR. For categorical data, number and percentage will be presented. For comparison of continuous data linear regression analyses or correlation (Spearman or Pearson) will used. For comparison of continuous data with categorical data logistic regression analysis will be used. For comparison of two sets of categorical data the chi-square test of Fisher's exact test will be utilized. For the radiological PFS analyses the estimates of the hazard ratio and corresponding 95% confidence interval will be tested using a Cox Proportional hazard model. For the overall survival, a stratified log-rank test will be used to compare between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥ 65 years with mCRPC previously treated with docetaxel
2. Medical or surgical castration with castrate level of testosterone (< 50 ng/dl) based on the EAU definition of castrate level of testosterone
3. Progressive disease according to PCWG2
4. Histologically proven prostate carcinoma
5. Health status allowing use of chemotherapy: G8 > 14; or G8 score ≤ 14 with geriatric assessment concluding to reversible impairment allowing use of chemotherapy
6. ECOG-PS 0, 1 or 2(ECOG-PS 2 should be related to prostate cancer)
7. Adequate hematologic, liver and renal functions:

   1. Neutrophil count ≥1.5 109/L
   2. Haemoglobin ≥10 g/ dL
   3. Platelet count ≥100.109/L
   4. Total bilirubin ≤ 1 the upper limit of normal (ULN)
   5. Transaminases ≤ 1.5 ULN
   6. Serum creatinine ≤ 2.0 ULN
8. Ongoing LHRH therapy at study entry
9. Signed informed consent

Exclusion Criteria:

1. History of severe hypersensitivity reaction (≥grade 3) to docetaxel
2. History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs
3. Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus)
4. Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments) (see Appendix E)
5. PS >2 not related to prostate cancer disease
6. G8 ≤ 14 with geriatric assessment contra-indicating standard cabazitaxel regimen
7. Concomitant vaccination with yellow fever vaccine
8. Patient who cannot be regularly followed or cannot answer to quality of life questionnaires because of psychological, social, familial or geographic reasons
9. Participation in another clinical trial with any investigational drug within 30 days prior to study enrolment.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 196 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Number of grade ≥ 3 neutropenia and/or neutropenic complications | Up to 11 months
  To evaluate the incidence of grade ≥ 3 neutropenia (measured at Day 7 and Day 14) and/or neutropenic complications (febrile neutropenia, neutropenic infection) with two schedules of cabazitaxel (bi-weekly versus tri-weekly) plus prednisone in elderly men (≥ 65 years) with mCRPC previously treated with a docetaxel-containing regimen.
  with two schedules of -+cabazitaxel (bi-weekly versus tri-weekly) plus prednisone in elderly men with mCRPC previously treated with a docetaxel-containing regimen

SECONDARY OUTCOMES:
Dose reductions | through study completion, an average of 40 weeks
  Up to 11 months
Radiological progression-free survival (rPFS) | Up to 11 months
  CT-Scan (abdominal/pelvic/chest) or whole body MRI and Bone scan
Time to PSA progression | Up to 11 months
  Assessed at C1D1, at every each subsequent visit and EOT
Time to first symptomatic Skeletal-Related Event (SRE) and incidence of SREs | Up to 11 months
  Assessed at C1D1, at every each subsequent visit and EOT
Time to opioid treatment (if relevant) | Up to 11 months
Prostate-specific antigen (PSA) response rate | Up to 11 months
  Assessed at C1D1, at every each subsequent visit and EOT
Quality of Life (FACT-P) | Up to 11 months
  Assessed at C1D1, at every each subsequent visit and EOT
Objective response rate (ORR) in measurable lesions (RECIST criteria 1.1 - only on metastasis | Up to 11 months
  CT-Scan (abdominal/pelvic/chest) or whole body MRI
Overall Survival (OS) | up to 11 months
Factors influencing survival | Up to 11 months
  Factors influencing survival (duration of response to first ADT, serum testosterone, cumulative dose of cabazitaxel, neutrophils/lymphocytes ratio, Gleason score, G8, grade ≥3 neutropenia)
Time to onset of grade ≥3 neutropenia | Up to 11 months
  Hematology every week until EOT
Grade ≥3 neutropenia duration ( from date of onset of grade ≥ 3 until grade ≤ 2) | Up to 11 months
  Hematology every week until EOT
Time to onset of grade ≥3 neutropenia by cycle | Up to 11 months
  Analysis of grade ≥3 neutropenia and/or neutropenia by cycle
Adverse events | Up to 11 months
Dose delay | Up to 11 months

OTHER OUTCOMES:
Proportion of patients achieving a best objective response of SD, PR or CR according to RECIST 1.1 specifically comparing those achieving >30% and >50% decrease in MDSC post-induction compared to those who did not achieve this reduction. | Up to 6 months
  Biomarker analysis
Proportion of patients achieving a >50% PSA response at 12 weeks and at any time specifically comparing those achieving >30% and >50% decrease in MDSC post-induction compared to those who did not achieve this reduction. | Up to 6 months
  Exploratory sub-study: biomarker analysis
Radiological progression-free survival (rPFS) according to PCWG2 criteria for all patients, in relation to percentage MDSC change (% maximum change and those achieving >30% and >50% decrease) | Up to 6 months
  Exploratory sub-study: biomarker analysis
Correlations between extent of MDSC (continuous) and NLR decline (continuous) | Up to 6 months
  Exploratory sub-study: biomarker analysis
Differences in peripheral blood immune populations (MDSCs, regulatory T-cells, T-effector and natural killer [NK] cells) with cabazitaxel responsiveness for Q2W and Q3W dosing schedule at week 6 and week 12 | Up to 6 months
  biomarkers analysis
  1. collection of blood (EDTA tube) at Baseline, C1D8,week 6, week 12 and EOT Collection of blood (RNA Paxgene): baseline
  2. platelet poor plasma isolation, PBMC isolation, PMN isolation and
  3. Flow cytometry assessments and FACS sorting Next-generation targeted sequencing of cfDNA RNA sequencing of baseline PaxGene
correlation between MDSC decline (>30% or >50%) with neutropenia (presence or absence) | Up to 6 months
  Hematology every week until EOT
  1. collection of blood (EDTA tube) at Baseline, C1D8,week 6, week 12 and EOT Collection of blood (RNA Paxgene): baseline
  2. platelet poor plasma isolation, PBMC isolation, PMN isolation and
  3. Flow cytometry assessments and FACS sorting Next-generation targeted sequencing of cfDNA RNA sequencing of baseline PaxGene
Associations between cabazitaxel dose, presence of neutropenia (C1D8), NLR conversion (wk6 and wk12) and MDSC decline (wk6 and wk12) | Up to 6 months
  biomarkers analysis
  1. collection of blood (EDTA tube) at Baseline, C1D8,week 6, week 12 and EOT Collection of blood (RNA Paxgene): baseline
  2. platelet poor plasma isolation, PBMC isolation, PMN isolation and
  3. Flow cytometry assessments and FACS sorting Next-generation targeted sequencing of cfDNA RNA sequencing of baseline PaxGene
To evaluate changes in peripheral blood immune populations at failure on cabazitaxel, with particular focus on CD38-positive MDSC subsets | Up to 6 months
  biomarkers analysis
  1. collection of blood (EDTA tube) at Baseline, C1D8,week 6, week 12 and EOT Collection of blood (RNA Paxgene): baseline
  2. platelet poor plasma isolation, PBMC isolation, PMN isolation and
  3. Flow cytometry assessments and FACS sorting Next-generation targeted sequencing of cfDNA RNA sequencing of baseline PaxGene
Associations between baseline MDSC and molecular underpinning (from cfDNA, specifically studying MYCN amplification and PTEN / TP53 aberration) | Up to 6 months
  biomarkers analysis
  1. collection of blood (EDTA tube) at Baseline, C1D8,week 6, week 12 and EOT Collection of blood (RNA Paxgene): baseline
  2. platelet poor plasma isolation, PBMC isolation, PMN isolation and
  3. Flow cytometry assessments and FACS sorting Next-generation targeted sequencing of cfDNA RNA sequencing of baseline PaxGene

CONTACTS AND LOCATIONS:
Overall Officials: Stephane OUDARD, MD, Ph.D, Principal Investigator — Hôpital Européen Georges Pompidou, Oncology Department
Locations (31):
- France (23):
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Saint André, CHU de Bordeaux, Bordeaux
  - Clinique Pasteur-CFRO, Brest
  - Centre Maurice Tubiana, Caen
  - Polyclinique Saint-Côme, Compiègne
  - CHU Henri-Mondor, Créteil
  - Clinique Victor Hugo, Le Mans
  - Centre Oscar Lambret Lille, Lille
  - Hôpital Belle-Isle, Metz
  - GHIRM, Montfermeil
  - Institut de Cancérologie du Gard - CHU, Nîmes
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Universitaire Tenon, Paris
  - Hôpital Cochin, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Rouen, Rouen
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - HIA Bégin 69 avenue de Paris, Saint-Mandé
  - Centre Hospitalier de Sens, Sens
  - Hôpitaux universitaires de Strasbourg, Strasbourg
  - Hôpital FOCH, Suresnes
  - Centre de cancérologie Les Dentellières, Valenciennes
- Germany (8):
  - Urologisch-onkologische Schwerpunktpraxis, Bernburg
  - Uniklinik Köln, Urologie, Uro-Onkologie, spezielle urologische und Roboter-assistierte Chirurgie, Cologne
  - Urologie und Kinderurologie Marienkrankenhaus Bergisch, Gladbach
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitäts-klinik für Urologie und Kinderurologie, Magdeburg
  - Urologische Praxis am Hasselbachplatz, Magdeburg
  - Universitätsklinikum Münster, Klinik für Urologie und Kinderurologie,, Münster
  - Studienpraxis Urologie, Nürtingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oudard S, Ratta R, Voog E, Barthelemy P, Thiery-Vuillemin A, Bennamoun M, Hasbini A, Aldabbagh K, Saldana C, Sevin E, Amela E, Von Amsberg G, Houede N, Besson D, Feyerabend S, Boegemann M, Pfister D, Schostak M, Huillard O, Di Fiore F, Quivy A, Lange C, Phan L, Belhouari H, Tran Y, Kotti S, Helissey C. Biweekly vs Triweekly Cabazitaxel in Older Patients With Metastatic Castration-Resistant Prostate Cancer: The CABASTY Phase 3 Randomized Clinical Trial. JAMA Oncol. 2023 Dec 1;9(12):1629-1638. doi: 10.1001/jamaoncol.2023.4255. PMID 37883073
- [Derived] Pobel C, Auclin E, Procureur A, Clement-Zhao A, Simonaggio A, Delanoy N, Vano YA, Thibault C, Oudard S. Cabazitaxel schedules in metastatic castration-resistant prostate cancer: a review. Future Oncol. 2021 Jan;17(1):91-102. doi: 10.2217/fon-2020-0672. Epub 2020 Dec 2. PMID 33463373